CLINICAL TRIAL: NCT05338320
Title: A Randomized Controlled Trial for Postoperative Analgesia in Patients Undergoing Elective Lumbar Fusion Operations Under General Anesthesia: Ultrasound Guided Erector Spinae Plane Block Versus Intrathecal Morphine
Brief Title: Postoperative Analgesia in Patients Undergoing Elective Lumbar Fusion Operations Under General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MD 102/2022
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General anesthesia and Ultrasound Guided Erector Spinae Plane Block (Active Comparator)
  Interventions: Procedure: Ultrasound Guided Erector Spinae Plane Block
- General anesthesia and intrathecal morphine (Active Comparator)
  Interventions: Drug: Intrathecal morphine
- General anesthesia using intravenous fentanyl (1µg/kg) (Other)
  Interventions: Other: General anesthesia using intravenous fentanyl (1µg/kg)

INTERVENTIONS:
Procedure: Ultrasound Guided Erector Spinae Plane Block — General anesthesia and Ultrasound Guided Erector Spinae Plane Block
  Arms: General anesthesia and Ultrasound Guided Erector Spinae Plane Block
Drug: Intrathecal morphine — General anesthesia and intrathecal morphine
  Arms: General anesthesia and intrathecal morphine
Other: General anesthesia using intravenous fentanyl (1µg/kg) — General anesthesia using intravenous fentanyl (1µg/kg)
  Arms: General anesthesia using intravenous fentanyl (1µg/kg)

SUMMARY:
It was proven that intrathecal opioids are considered as an effective means of pain control in several major surgical interventions including spine surgeries. Intrathecal morphine added to a spinal anesthesia reduces acute pain after spine surgeries but has side effects, including dose dependent respiratory depression, nausea, vomiting, pruritus, and sedation. Ultrasound guided Erector Spinae Plane Block (ESPB) was first described in 2016.Recent case reports suggest a positive effect of ultrasound guided ESPB on pain for multiple indications including lumbar spine fusion and scoliosis surgery, with a very low risk of complications as there are no structures in close proximity at risk of needle injury.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 25 to 35 kg/m².
* American Society of Anesthesiologist (ASA) physical status I or II.

Exclusion Criteria:

* patient's refusal
* Altered mental status
* Known allergy to study drugs (bupivacaine or morphine)
* Local infection at site of puncture.
* Known case with any pulmonary disease
* Known case with Obstructive sleep apnea (OSA)
* Coagulopathy and /or thrombocytopenia
* Severe hepatic or kidney impairment

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Time to first requested rescue analgesia (Minutes). | First 24 hours after surgery.
  Time to first requested rescue analgesia (Minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt